CLINICAL TRIAL: NCT06856109
Title: 68Ga-Pentikra PET/CT Imaging Study in Healthy Subjects
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: KY20252025
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- healthy volunteers (Experimental): Ten normal volunteers were recruited to perform 68Ga-Pentikra PET/CT imaging to assess the safety, biodistribution and radiation dosimetry of 68Ga-Pentikra.
  Interventions: Diagnostic Test: 68Ga-Pentikra PET/CT Scan

INTERVENTIONS:
Diagnostic Test: 68Ga-Pentikra PET/CT Scan — 68Ga-Pentikra Injection, Intravenous, administered at 0.05 mCi/kg by weight.

SUMMARY:
This is a prospective, interventional clinical pilot study that recruited 10 normal volunteers who underwent 68Ga-Pentikra PET/CT imaging to evaluate the safety, biodistribution and radiation dosimetry of 68Ga-Pentikra in normal volunteers.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age: 18 ~ 60 years old (including boundary values); 2) Gender: male or female; 3) Body weight: males weighing ≥50kg, females weighing ≥45kg, and body mass index [BMI = weight (kg)/height 2 (m2)] within the range of 19.0 ~ 26.0kg/m2 (including boundary values); (4) Subjects can fully understand and voluntarily participate in this experiment, and sign the informed consent form.

Exclusion Criteria:

- 1) Minors, pregnant women, lactating women, and those with severe hepatic or renal insufficiency (alanine aminotransferase exceeding the upper limit of normal values by 8-10 times and serum creatinine of 186-442 umol/L).

2) Previous history of tumour and surgery; 3) Other conditions judged by the investigator to be unsuitable as study subjects .

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Standardized uptake value | 1 day from injection of the tracer
  68Maximum standardised uptake values of Ga-Pentikra in regions of interest (ROIs) of the heart, lungs, liver, kidneys, spleen and brain in healthy subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine,Xijing Hospital, Fourth Military Medical University, Xi'an, China, Xi'an, Shaanxi Province, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No